CLINICAL TRIAL: NCT06110546
Title: Impact of Methadone on Prolonged Mechanical Ventilation in Patients on Continuous Treatment With Opioids, a Randomized Trial (IMPACTOR Study)
Brief Title: Impact of Methadone on Prolonged Mechanical Ventilation in Patients on Continuous Treatment With Opioids
Acronym: IMPACTOR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: very low recruitment
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Pascal Kingah, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HSC-MS-22-0689
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Results first posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Effect of Methadone on the Duration on Mechanical Ventilation
Keywords: opioids; mechanical ventilation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methadone group (Experimental)
  Interventions: Drug: Methadone group
- Non-Methadone group (Active Comparator)
  Interventions: Drug: Usual care

INTERVENTIONS:
Drug: Methadone group — Participants will be started on Methadone 5mg, 10mg or 15mg every 8 hours depending on Fentanyl drip rate (0-100mcg/hr, 100-200mcg/hr or >200mcg/hr) or hydromorphone drip rate (0-1.5mg/hr, 1.5-3mg/hr, or >3mg/hr).
  Arms: Methadone group
Drug: Usual care — Participants will receive usual care with IV Fentanyl or hydromorphone per hospital protocols
  Arms: Non-Methadone group

SUMMARY:
The purpose of this study is to determine the effect of methadone on the duration on mechanical ventilation in critically ill patients receiving more than 72 hours of mechanical ventilation (MV) by comparing the number of ventilator free days from enrollment to the time of discharge, to assess the safety of methadone administration in critically ill patients while in the hospital and to determine hospital length of stay from the time of enrollment to the time of discharge

ELIGIBILITY:
Inclusion Criteria:

* Patients on Intermittent mandatory ventilation (IMV) for more than 72 hours
* Patients infused Fentanyl or Hydromorphone for more than 72 hours
* Patients with evidence of reversal of process that caused respiratory failure, adequate oxygenation (PaO2/fraction of inspired oxygen (FiO2)>200; Positive end expiratory pressure (PEEP)≤8 and Ph≥7.2
* Patients hemodynamically stable
* Patients with a failed single or multiple attempts at spontaneous breathing trials

Exclusion Criteria:

* Patients with history of opioid drug abuse
* Patients receiving schedule II narcotics on a chronic basis for longer than 6 months prior to ICU admission or on other analgesic infusions other than Fentanyl or Hydromorphone
* Patients with cervical spinal cord injury or neuromuscular disease
* Patients with end stage liver disease at ICU admission (ie, International normalized ratio ≥2and not taking warfarin and/or a total serum bilirubin ≥1.5 times above normal limits
* Patients with prolonged QTc interval ≥500
* Patients with prior history of cardiac conduction defects or sudden death
* Patients with QTc increase of ≥60 milliseconds above the value of prior EKGs measured during current ICU admission
* Patients with more than 5 days on IV analgesia
* Patients intubated for more than 3 days
* Patients without feeding tubes
* Patients not receiving enteral feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2024-02-18 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pascal Kingah, MD,MPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 2 participants enrolled, 1 withdrew before randomization.
Period: Overall Study
Arm/Group | Methadone Group | Non-Methadone Group
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Includes all participants that were randomized. 0 participants were randomized to the non-methadone group arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Methadone Group | Non-Methadone Group | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 1 |  | 1
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 |  | 1
  Male | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 1 |  | 1
  White | 0 |  | 0
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1
Cause of Lung Injury [Count of Participants; unit: Participants]
  Pneumonia | 1 |  | 1
  Aspiration | 0 |  | 0
  Non-pulmonary Sepsis | 0 |  | 0
  Chronic Obstructive Pulmonary Disease (COPD) Exacerbation | 0 |  | 0
  Other Causes | 0 |  | 0
Weight [Mean (Standard Deviation); unit: Kilograms] | 129.9 |  | 129.9
Duration on ventilator at time of randomization [Mean (Standard Deviation); unit: hours] | 78 |  | 78

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants on Methadone That Get Extubated
Time Frame: from day of intubation to day 5
Population: 0 participants were randomized to the non-methadone group arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Methadone Group | Non-Methadone Group
Number analyzed (Participants) | 1 | 0
Participants | 1 |

2. Secondary Outcome: Number of Participants That Develop Prolonged Corrected QT Interval (QTC) After Administration of Methadone
Time Frame: from first day patient given Methadone to date patient discharged or transferred from hospital (up to about 27 days after admission)
Population: 0 participants were randomized to the non-methadone group arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Methadone Group | Non-Methadone Group
Number analyzed (Participants) | 1 | 0
Participants | 0 |

3. Secondary Outcome: ICU Length of Stay
Time Frame: From time of admission to ICU to time of discharge from ICU (about 27 days after admission)
Population: 0 participants were randomized to the non-methadone group arm.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Methadone Group | Non-Methadone Group
Number analyzed (Participants) | 1 | 0
days | 27 |

4. Secondary Outcome: ICU Mortality
Time Frame: end of ICU stay (up to about 27 days after admission)
Population: 0 participants were randomized to the non-methadone group arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Methadone Group | Non-Methadone Group
Number analyzed (Participants) | 1 | 0
Participants | 0 |

5. Secondary Outcome: Hospital Length of Stay
Time Frame: from time to admission to time of discharge from hospital (about 27 days after admission)
Population: 0 participants were randomized to the non-methadone group arm.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Methadone Group | Non-Methadone Group
Number analyzed (Participants) | 1 | 0
days | 27 |

6. Secondary Outcome: Hospital Mortality.
Time Frame: end of hospital stay (up to about 27 days after admission )
Population: 0 participants were randomized to the non-methadone group arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Methadone Group | Non-Methadone Group
Number analyzed (Participants) | 1 | 0
Participants | 0 |

ADVERSE EVENTS:
Time Frame: 27 days
Description: 0 participants are at risk for serious adverse events, all cause mortality and other (not including serious) adverse events because 0 participants were enrolled in the Non-Methadone Group arm.
Arm/Group | Methadone Group | Non-Methadone Group
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-05): https://cdn.clinicaltrials.gov/large-docs/46/NCT06110546/Prot_SAP_000.pdf